CLINICAL TRIAL: NCT05397236
Title: A Comparative Study Between the Effect of Addition of MgSO4 or Dexamethasone to Bupivacaine on the Prolongation of Ultrasound-guided Quadratus Lumboram Block
Brief Title: Addition of MgSO4 or Dexamethasone to Bupivacaine on the Prolongation of Ultrasound-guided Quadratus Lumboram Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada M.Samir, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 256/2021
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine Magnesium sulphate group (Active Comparator): Patients received QL block with 20 ml of 0.25% bupivacaine (2, 4)plus 5 ml of 10% MgSO4.
  Interventions: Drug: Bupivacaine- Magnesium
- Bupivacaine Dexamethasone group (Active Comparator): Patients received QL block with 20 ml of 0.25% bupivacaine (2,4)plus 2 ml of 8 mg dexamethasone plus 3 ml of 0.9% NS.
  Interventions: Drug: Bupivacaine dexamethasone
- bupivacaine saline group (Active Comparator): Patients received QL block with 20 ml of 0.25% bupivacaine (2,4)plus 5 ml of 0.9% NS.
  Interventions: Drug: Bupivacaine saline

INTERVENTIONS:
Drug: Bupivacaine- Magnesium — Patients received QL block with 20 ml of 0.25% bupivacaine (2, 4)plus 5 ml of 10% MgSO4.
  Arms: Bupivacaine Magnesium sulphate group
Drug: Bupivacaine dexamethasone — Patients received QL block with 20 ml of 0.25% bupivacaine (2,4)plus 2 ml of 8 mg dexamethasone plus 3 ml of 0.9% NS.
  Arms: Bupivacaine Dexamethasone group
Drug: Bupivacaine saline — Patients received QL block with 20 ml of 0.25% bupivacaine (2,4)plus 5 ml of 0.9% NS.
  Arms: bupivacaine saline group

SUMMARY:
The goal of postoperative pain management is the provision of comfort, early mobilization and improved respiratory function without causing inadequate sedation and respiratory compromise, which can be achieved through using regional anethesia.

This study aimed to assess the analgesic effect of adding dexamethasone or magnesium sulphate with bupivacaine in ultrasound-guided QLB to prolong its duration in patients undergoing open abdominal surgeries in the early postoperative period regarding pain relief After approval of the ethical committees in Ain Shams University Hospitals, patients undergoing open abdominal surgeries were included in the study, and were divided into three groups (n=22; each); group M, D and group C. In Group A, patients (n=22) received 20 ml bupivacaine 0.25% plus 5 ml of 10% MgSO. In group B, patients (n=22) received 20 ml bupivacaine 0.25% plus 8 mg dexamethasone (2 ml) plus 3 ml 0.9% NaCl. In group C (control), patients (n=22) received 20 ml bupivacaine plus 5 ml 0.9% NaCl.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II
* aged 18 to 65 years
* body weight ≥ 60 kg and ≤ 90 kg
* scheduled for open abdominal surgeries

Exclusion Criteria:

* Patients' refusal to participate in the study
* history of allergy to the medications used in the study
* hepatic disease
* renal disease
* known neurologic disorders
* psychiatric disorder
* chronic treatment with calcium channel blockers
* hyper-magnesemia
* coagulopathy
* anatomical abnormalities
* hemodynamic instability
* local infection
* suspected intra- abdominal sepsis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Duration of post-operative analgesia | 24hours
  Time from completion of the block to the first request of rescue analgesia.

SECONDARY OUTCOMES:
Mean arterial blood pressure | 24 hours
  Measured before induction of anesthesia (base line), upon arrival to the PACU, after 30 and 60 min. If hypotension (MBP < 20% of the base line value) occurred, 3 mg increments of ephedrine repeated every 5 min if required was given. MBP was then recorded at 2, 6, 12 and 24 post-operative hours.
Heart rate | 24 hours
  Recorded before induction of anesthesia (base line),upon arrival to the PACU, after 30 and 60 min. If bradycardia (HR <50 bpm) occurred, 0.5 mg atropine was given. HR was then recorded at 2, 6, 12 and 24 post-operative hours.
The severity of post-operative pain at rest | 24 hours
  By using the Visual Analogue Scale (VAS); from 0= no pain, to 10=worst imaginable pain. Assessed upon arrival to the PACU, after 30 and 60 min. The VAS was then recorded at 2, 4, 6, 8, 12 and 24 post-operative hours.
The severity of post-operative pain with movement (bilateral knee flexion) | 24 hours
  By using the Visual Analogue Scale (VAS); from 0= no pain, to 10=worst imaginable pain. Assessed at 2, 4, 6, 8, 12 and 24 post-operative hours
Number of patients requiring post-operative rescue analgesia | 24 hours
  Number of patients requiring pethidine in the 24 hours post-operative period
Total dose of pethidine given | 24 hours
  The cumulative total pethidine doses given to each patient in the 24 hours post-operative period.
Occurrence of nausea and/or vomiting: | 24 hours
  Number of patients who develop nausea and/or vomitting
Time to first ambulation | 24 hours
  The time to the start of movement by each patient in the 24 hours post-operative period
The analgesic satisfaction at 24 post-operative hours | 24 hours
  Patients were asked to report their satisfaction with the pain management; assessed as, 1 = poor, 2 = fair, 3 = good, and 4 = excellent.
Inadvertent femoral nerve block | 24 hours
  number of patients who develop lower limb weakness
Local Anesthetic Systemic Toxicity (LAST): | 24 hours
  As any regional anesthesia technique with local anesthetic is associated with potential systemic absorption of local anesthetics.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No